CLINICAL TRIAL: NCT00835224
Title: Safety and Efficacy of L-NAME and Midodrine to Increase MAP in Persons With Tetraplegia
Brief Title: Safety and Efficacy of L-NAME and Midodrine to Increase MAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A6161-W; VA Project #5481-08-017 (Other: JJP VAMC RR&D)
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Orthostatic Hypotension; Spinal Cord Injury
Keywords: Spinal Cord Injury; Orthostatic Hypotension; Blood Pressure; Midodrine Hydrochloride; L-NAME
MeSH Terms: conditions — Hypotension, Orthostatic; Spinal Cord Injuries | interventions — NG-Nitroarginine Methyl Ester; Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Midodrine (Experimental): A drug to treat low blood pressure.
  Interventions: Drug: Midodrine
- L-Name (Experimental): L-Name: A non-selective inhibitor of nitric oxide synthase and placebo. It has been used experimentally to induce hypertension.
  Interventions: Drug: L-NAME
- Placebo (Placebo Comparator): Placebo: A pill with an inactive substance that looks like the study drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-NAME — A non-selective inhibitor of nitric oxide synthase and placebo. It has been used experimentally to induce hypertension.
  Arms: L-Name
Drug: Midodrine — To treat low blood pressure.
  Arms: Midodrine
Drug: Placebo — A pill with an inactive substance that looks like the study drug.
  Arms: Placebo

SUMMARY:
After a spinal cord injury the brain is no longer completely in control of the body below the level of injury. This affects many organs and systems in the body, we are interested in understanding how a spinal cord injury affects blood pressure and blood flow to the brain. We are going to study blood pressure while the person is seated in a wheelchair before and after we give the subject medications which should increase blood pressure in a laboratory setting and over the course of a normal day in persons with spinal cord injury.

DETAILED DESCRIPTION:
Blood pressure regulation is compromised in persons with tetraplegia due to de-centralization of sympathetic cardiovascular control, associated with hypotension during upright positioning (7, 10, 18, 33). An alpha receptor agonist (midodrine hydrochloride) has been reported to raise blood pressure in persons with tetraplegia (25, 26, 30). Midodrine is the only drug that is presently available to treat orthostatic hypotension. In the clinical armamentarium, it is always beneficial to have agents from multiple drug classes to treat a condition. In the treatment of hypertension, several classes of drugs may be prescribed to lower blood pressure, alone or in combination. The clinician and patient would benefit if another class of drug, with a totally separate mechanism of action, were available to treat orthostatic hypotension. A nitric oxide synthase inhibitor (NOSi), nitro-L-arginine methyl ester (L-NAME), has been shown by our group to "normalize" blood pressure in persons with tetraplegia (32). The safety and efficacy of these two hypertensive agents has not been investigated or compared in persons with chronic tetraplegia. Although the mechanism of action of each of these agents is appreciated, the relative cardiovascular effect in persons with SCI compared with controls is not known. The study will determine the efficacy and safety of these two medications at restoring mean arterial pressure (MAP) during daily activities in persons with chronic tetraplegia. Furthermore, the implication of restoring MAP to normal levels (80 10 mmHg) in individuals with tetraplegia on cardiovascular, autonomic, hormonal and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

Spinal Cord Injured Subjects:

* chronic spinal cord injury (1 year post injury) with a seated MAP of 65mmHg (almost all individuals with tetraplegia demonstrate this)
* Male or female with an age of 18 - 65 years

Control Subjects:

* Male or female with an age of 18 - 65 years

Exclusion Criteria:

Spinal Cord Injured Subjects:

* acute illness
* cardiovascular disease
* renal disease
* medications that affect the cardiovascular system

Control Subjects:

* acute illness
* cardiovascular disease
* renal disease
* medications that affect the cardiovascular system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Wecht, EdD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States

REFERENCES:
- [Result] Wecht JM, Radulovic M, Rosado-Rivera D, Zhang RL, LaFountaine MF, Bauman WA. Orthostatic effects of midodrine versus L-NAME on cerebral blood flow and the renin-angiotensin-aldosterone system in tetraplegia. Arch Phys Med Rehabil. 2011 Nov;92(11):1789-95. doi: 10.1016/j.apmr.2011.03.022. Epub 2011 Jul 16. PMID 21762873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 34 subjects were consented 24 completed testing. Subjects were recruited through the Center of Excellence for the Medical Consequences of Spinal Cord Injury (SCI) from June 2010 to August of 2013.
Pre-assignment Details: Eligibility criteria were covered by the study coordinator prior to enrollment.
Groups:
- All Participants: All Participants visited the laboratory on 3 occasions for a 4-5 hour observation of blood pressure following administration of a non-selective inhibitor of nitric oxide synthase (L-NAME) an alpha-agonist (midodrine) or placebo. The interventions were administered in random order on separate laboratory visits.
Period: Overall Study
Arm/Group | All Participants
Started | 34
Completed | 24
Not Completed | 10

BASELINE CHARACTERISTICS:
Population: 30 subjects were anticipated but 34 were enrolled following an IRB approval to expand the n. Increased recruitment was due to a number of subjects withdrawing from participation for various reasons listed below.
Groups:
- All Participants: All participants were studied on three laboratory visits and underwent seated blood pressure assessment before and after administration of Midodrine, L-NAME or placebo, which were given in random order.
Arm/Group | All Participants
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Time Frame: Blood pressure during the 4 hour period after no drug, L-NAME (IV: 1.0 mg/kg) and midodrine (PO: 10.0 mg) administration
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Arm 1A: Spinal Cord Injured participants - Seated blood pressure after administration of a nitric oxide synthase inhibitor (L-NAME)over the course of 3 hours
- Arm 1B: Non disabled participants seated systolic blood pressure for 3 hours after administration of a nitric oxide synthase inhibitor (L-NAME)
- Arm 2A: Spinal cord injured participants seated systolic Blood Pressure for 3 hours after administration of midodrine or
- Arm 2B: Non disabled participants seated systolic blood pressure for 3 hours after administration of midodrine.
- Arm 3A: Spinal cord injured participants systolic blood pressure for 3 hours after administration of no drug
- Arm 3B: Non disabled participants seated systolic blood pressure for 3 hours after administration of no drug.
Arm/Group | Arm 1A | Arm 1B | Arm 2A | Arm 2B | Arm 3A | Arm 3B
Number analyzed (Participants) | 15 | 10 | 15 | 10 | 15 | 10
mmHg | 120 (17) | 112 (10) | 117 (19) | 109 (5) | 96 (12) | 109 (6)

ADVERSE EVENTS:
Arm/Group | Arm 1A | Arm 1B | Arm 2A | Arm 2B | Arm 3A | Arm 3B
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/9 | 0/15 | 0/9 | 0/15 | 0/9
Other Adverse Events (participants affected / at risk) | 0/15 | 0/9 | 0/15 | 0/9 | 0/15 | 0/9

LIMITATIONS AND CAVEATS:
Study population was relatively small and were not blinded to the interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No